CLINICAL TRIAL: NCT00834691
Title: Anemia in Chronic Heart Failure: Etiology, Comparisons With Renal Disease, and Relationships With Biomarkers and Left Ventricular Remodeling.
Brief Title: An Evaluation of the Causes of Anemia in Patients With Heart Failure
Acronym: ANCHOR
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Eileen O'Meara, Montreal Heart Institute
Other Study IDs: 07-938
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: Anemia; Heart Failure; Chronic Renal Failure
Keywords: Inflammation; Oxidative stress; Estimated glomerular filtration rate
MeSH Terms: conditions — Anemia; Heart Failure; Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum samples for analysis of biomarkers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients with anemia and systolic heart failure
- 2: Patients with systolic heart failure but without anemia
- 3: Patients with at least moderate chronic renal failure, with or without anemia and without systolic heart failure.

SUMMARY:
Anemia is frequent in patients with heart failure. Few studies have clearly addressed the causes of anemia in patients with HF. The purpose of this study is to evaluate differences in blood concentrations of various substances related to inflammation, oxidative stress, renal function and other processes between individuals with 1) heart failure and anemia, 2) heart failure without anemia and 3) patients with kidney disease without systolic heart failure. This study will help to better understand the reasons why some people with heart failure have anemia.

ELIGIBILITY:
Inclusion Criteria:

Groups 1 and 2

* Age >18 years
* Group 1: hemoglobin < 120g/L in women and < 130 g/L in men (in agreement with the WHO definition of anemia)
* Group 2: hemoglobin > or = 120g/L in women and > or = 130 g/L in men
* Patients with chronic HF referred to a specialized HF clinic, or with a diagnosis of HF at least 6 months prior to enrolment
* NYHA functional class II-IV at the time of enrolment
* Patients already on CHF medical therapy (ACEI or ARBs, beta-blockers if tolerated, with or without digoxin, and loop diuretics), at stable doses for > or = 1 month
* LVEF < or = 40% within 6 months prior to patient enrolment, by echocardiography, radionuclide ventriculography or perfusion scan, or radiologic angiography

Inclusion criteria - group 3

* Age >18 years
* At least moderate CRF (eGFR < 60ml/min/1,73m2)
* With or without anemia
* LVEF > or = 50% within 6 months prior to patient enrolment, by echocardiography, radionuclide ventriculography or perfusion scan, or radiologic angiography

Exclusion Criteria (all groups):

* Recent acute renal failure episode (< 1 month)
* Red blood cells (or other blood component) transfusions or EPO therapy within 3 months prior to enrolment
* Iron, B12 or folic acid supplements used to treat anemia (< 3 months)
* Evidence of active GI bleeding
* Recent acute coronary syndrome or decompensated HF episode (< 1 month)
* Complex congenital heart disease
* Known malignant hematologic or other active neoplasia
* Immunosuppressive therapy, chemotherapy or radiotherapy within 3 months prior to enrolment
* Recent acute decompensation of a chronic inflammatory disease (e.g. chronic inflammatory bowel disease, rheumatoid arthritis, collagen vascular disease) within 3 months prior to enrolment
* Recent viral or bacterial syndrome (< 2 weeks)
* Active or recent viral hepatitis (< 3 months)
* Pregnant women
* Potential for non compliance to tests involved in this protocol
* Incapacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and eighty (180) patients will be enrolled in three groups.
  Group 1: This group will involve 80 patients with anemia (hemoglobin < 120g/L in women and < 130 g/L in) and systolic heart failure (LVEF < or = 40%; New York Heart Association -NYHA- functionnal class II-IV).
  Group 2: This group will include 50 patients with systolic heart failure (LVEF < or = 40%; New York Heart Association -NYHA- functionnal class II-IV), but without anemia (hemoglobin > or = 120g/L in women and > or = 130 g/L in men).
  Group 3 : 50 patients with at least moderate CRF (eGFR < 60ml/min/1,73m2), and LVEF > or = 50%, with or without anemia.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
TNF alpha concentrations | Visit 2 (within 2 weeks of baseline visit)

SECONDARY OUTCOMES:
Various echocardiographic measurements, markers of inflammation, oxydative stress, neurohormonal activity and myocardial extracellular matrix turnover will be measured | Visit 2 (within 2 weeks of baseline visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] O'Meara E, Clayton T, McEntegart MB, McMurray JJ, Lang CC, Roger SD, Young JB, Solomon SD, Granger CB, Ostergren J, Olofsson B, Michelson EL, Pocock S, Yusuf S, Swedberg K, Pfeffer MA; CHARM Committees and Investigators. Clinical correlates and consequences of anemia in a broad spectrum of patients with heart failure: results of the Candesartan in Heart Failure: Assessment of Reduction in Mortality and Morbidity (CHARM) Program. Circulation. 2006 Feb 21;113(7):986-94. doi: 10.1161/CIRCULATIONAHA.105.582577. Epub 2006 Feb 13. PMID 16476847
- [Background] de Denus S, Tardif JC, White M, Bourassa MG, Racine N, Levesque S, Ducharme A. Temporal variations in hematocrit values in patients with left ventricular dysfunction: Relationship with cause-specific mortality and morbidity and optimal monitoring--further insights from SOLVD. Can J Cardiol. 2008 Jan;24(1):45-8. doi: 10.1016/s0828-282x(08)70547-6. PMID 18209768
- [Derived] O'Meara E, Rouleau JL, White M, Roy K, Blondeau L, Ducharme A, Neagoe PE, Sirois MG, Lavoie J, Racine N, Liszkowski M, Madore F, Tardif JC, de Denus S; ANCHOR Investigators. Heart failure with anemia: novel findings on the roles of renal disease, interleukins, and specific left ventricular remodeling processes. Circ Heart Fail. 2014 Sep;7(5):773-81. doi: 10.1161/CIRCHEARTFAILURE.114.001100. Epub 2014 Jul 15. PMID 25027873